CLINICAL TRIAL: NCT06198894
Title: Study on the Efficacy of in Office Steroid-eluting Sinus Stent Implantation in Chronic Rhinosinusitis Patients With Uncontrolled Postoperative Symptoms
Brief Title: Steroid-eluting Sinus Stent for Chronic Rhinosinusitis Patients With Uncontrolled Postoperative Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng Liu (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery; Deputy Dean of Tongji Medical College; Deputy Dean of Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stent-001
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Chronic Sinusitis
Keywords: steroid-eluting sinus stent; mucous edema
MeSH Terms: interventions — Methylprednisolone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Stent-001 is a randomized (1:1), sham-controlled, parallel group, single-blind, non-inferiority, multicenter study
Who Masked: Participant
Masking Description: Participants were blindfolded and earmuffed during the baseline procedure and follow-up endoscopic examinations. Implants were biodegradation at Week 4 to allow blinded assessment of bilateral edema score grade.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid-eluting Sinus Implant (Experimental): In-office bilateral placement of the sinus stent; Systemic glucocorticoid placebo; saline irrigations (250ml) twice daily
  Interventions: Procedure: steroid-eluting sinus stent implant; Drug: saline irrigations; Drug: Placebo
- Control (Sham Comparator): In-office bilateral sham procedure; Systemic glucocorticoid; saline irrigations (250ml) twice daily
  Interventions: Drug: Systemic glucocorticoids; Drug: saline irrigations; Procedure: sham procedure

INTERVENTIONS:
Procedure: steroid-eluting sinus stent implant — In-office bilateral placement of the steroid-eluting sinus stent in the ethmoid sinuses under local anesthesia
  Other Names: BISORB bioabsorbable steroid-eluting sinus stent
  Arms: Steroid-eluting Sinus Implant
Drug: Systemic glucocorticoids — Groups were given oral methylprednisolone (32 mg/d on days 1-5; 16 mg/d on days 6-10; and 8 mg/d on days 11-20),
  Other Names: Medrol
  Arms: Control
Drug: saline irrigations — Patients were routinely treated with saline irrigations (250ml) twice daily
  Other Names: 0.9% sodium chloride solution
Drug: Placebo — Groups were given systemic glucocorticoid placebo
  Other Names: Systemic glucocorticoid placebo
  Arms: Steroid-eluting Sinus Implant
Procedure: sham procedure — The sham procedure was performed in-office under local anesthesia
  Other Names: In-office bilateral sham procedure of stent placement
  Arms: Control

SUMMARY:
Stent-001 study is a randomized controlled clinical trial with the steroid-eluting Sinus in 96 chronic rhinosinusitis patients with uncontrolled postoperative symptoms

DETAILED DESCRIPTION:
Stent-001 is a randomized (1:1), sham-controlled, parallel group, single-blind, non-inferiority, multicenter study in 96 chronic rhinosinusitis patients who had prior endoscopic sinus surgery and presented with uncontrolled postoperative symptoms. The objective was to evaluate the safety and clinical efficacy of sinus stents relative to systemic glucocorticoids. The steroid-eluting sinus stent consist of a bioabsorbable self-expanding sinus implant coated with 625 mcg of mometasone furoate (MF) and a single-use delivery system. Implant is placed in-office in the ethmoid sinus under local anesthesia. The coating on the sinus stent implant provides controlled release of MF to the sinus mucosa over 30 days.

ELIGIBILITY:
Inclusion Criteria:

* The patient underwent pre-functional endoscopic sinus surgery and bilateral ethmoidectomy (for at least 3 months), and was identified by the clinician as having uncontrolled symptoms (Diagnostic criteria of EPOS 2020) with a Snot-22 score of at least 20;
* Edema score of bilateral nasal endoscopy was 2 points both;
* Understands the purpose and procedures of the trial and voluntarily signs the informed consent form;
* The female subjects had no pregnancy or lactation plans during the treatment and follow-up period;
* The subject has not participated in other clinical trials in the previous three months and agrees not to participate in other clinical trials until the end point of this trial was reached;
* Subjects were 18-65 years old, male or non-pregnant women;

Exclusion Criteria:

* Grade 2 or more nasal polyp scores in either nasal cavity (i.e., polyps extending beyond the middle nasal passage)
* The subject has a known allergic reaction or contraindication to the device material and its degradation products (mamethasone citrate, L-polylactic acid, racemic polylactic acid, lactide lactate, lactic acid);
* Subjects had cystic fibrosis, congenital ciliary dyskinesia, fungal globular sinusitis, systemic vasculitis and granulomatous diseases, tumors, and immune deficiency.
* The patient underwent endoscopic nasal surgery within 3 months.
* Acute exacerbation of allergic rhinitis, acute exacerbation of CRS, upper respiratory tract infection, or common cold in the 4 weeks prior to screening visit;
* Have a clinically serious metabolic, cardiovascular, immune, neurological, blood, digestive, cerebrovascular, or respiratory disease, or any condition that the investigator believes interferes with the evaluation of the study results or affects the safety of the subjects;
* Symptomatic seasonal allergic rhinitis, and/or, depending on the season, expected to develop symptoms and require nasal spray hormone therapy within 4 weeks of randomization,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Sino-Nasal Outcome Test Scores (SNOT-22) | Change from Baseline to Week 4
  The change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment between the two arms was measured. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis is by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT includes 22 questions (symptoms and social/emotional consequences of rhinosinusitis), each of which are rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores representing worse outcome.

SECONDARY OUTCOMES:
Change in Sino-Nasal Outcome Test Scores (SNOT-22) | Change from Baseline to Week 1, 2, 8, 12
  The change in Sino-Nasal Outcome Test scores (SNOT-22) scores pre- and post-treatment between the two arms was measured. The Sino-Nasal Outcome Test asks subjects to rate how "bad" their rhinosinusitis is by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT includes 22 questions (symptoms and social/emotional consequences of rhinosinusitis), each of which are rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores representing worse outcome.
Change in nasal symptoms | Change from Baseline to Week 1, 2, 4, 8, 12
  Nasal symptoms measured by Visual analog score. The four nasal symptoms (nasal obstruction, rhinorrhea, headache and olfactory disorder) involved in assigning the total nasal symptom score(TNSS). The symptoms are graded on a10-point scale (0 = no symptoms;10 = most severe symptoms).
Rescue medication use | Week 4 and Week 12
  If polyps and/or the moderate to severe clinical symptoms of CRS were relapsed and/or not controlled throughout the study period, rescue medication of corticosteroids for the experimental group will be used and recorded.
The rate of surgery rate | Week 4 and Week 12
  The rate of nasal endoscopic surgery for the experimental or control group throughout the study period will be recorded.
Lund-Kennedy Scoring for Nasal Endoscopy | Change from Baseline to Week 1, 2, 4
  The Lund Kennedy scoring system for nasal endoscopy rates the severity of the sinusitis based on the endoscopic appearance of the nasal mucosa. Edema, secretions, and the presence of polyps are rated from 0-2, for a total maximum score of 6 per each side of the nose. Higher scores represent more severe disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Forwith KD, Han JK, Stolovitzky JP, Yen DM, Chandra RK, Karanfilov B, Matheny KE, Stambaugh JW, Gawlicka AK. RESOLVE: bioabsorbable steroid-eluting sinus implants for in-office treatment of recurrent sinonasal polyposis after sinus surgery: 6-month outcomes from a randomized, controlled, blinded study. Int Forum Allergy Rhinol. 2016 Jun;6(6):573-81. doi: 10.1002/alr.21741. Epub 2016 Mar 14. PMID 26992115
- [Background] Van Zele T, Gevaert P, Holtappels G, Beule A, Wormald PJ, Mayr S, Hens G, Hellings P, Ebbens FA, Fokkens W, Van Cauwenberge P, Bachert C. Oral steroids and doxycycline: two different approaches to treat nasal polyps. J Allergy Clin Immunol. 2010 May;125(5):1069-1076.e4. doi: 10.1016/j.jaci.2010.02.020. PMID 20451040